CLINICAL TRIAL: NCT02994810
Title: Orientation Effects of Breastfeeding for Mothers in a Private Hospital: Randomized Controlled Trial
Brief Title: Orientation Effects of Breastfeeding for Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Salete Matos, Principal Investigator, Hospital Moinhos de Vento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMV - Breastfeeding
Record Dates: First submitted 2016-01-07; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Orientation
MeSH Terms: conditions — Breast Feeding; Orientation, Spatial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Guidelines and review of the breastfeeding techniques.
  Interventions: Other: Breastfeeding guidance
- Control group (No Intervention): The control group will receive home visits only when the baby is 6 months of life, they will be re-evaluated by the researchers as the practice of exclusive breastfeeding and the technical and nursing management, and will be asked about the main difficulties encountered in maintaining breastfeeding.

INTERVENTIONS:
Other: Breastfeeding guidance — Breastfeeding guidance
  Arms: Intervention group

SUMMARY:
The benefits of breastfeeding are increasingly known of the population and breastfeeding rates in the country have been increasing, but still are below satisfactory to the Ministry of Health (MH) and the World Health Organization (WHO).

Simple Strategies to guide and support the mother contributes to increasing knowledge about breastfeeding and can have positive impacts on breastfeeding rates.

DETAILED DESCRIPTION:
Assess the impact of guidance on breastfeeding duration of exclusive breastfeeding in the first six months of a baby's life.

110 pairs of mother / baby - Recruitment: Private Hospital of Porto Alegre.

The first stage was carried out in the maternity - Orientation: Breastfeeding Importance Handle Correct, Positioning mother and baby, socioeconomic data and demographics. For the intervention group held three home visits:

10th day, 1st and 2nd month of the baby's life. At 6 months were made telephone contact for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Mothers living in the city of Porto Alegre

Exclusion Criteria:

* Mothers who test positive for HIV, poor hearing, visual and mental disorders, preterm infants, twin hospitalized

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Effects of Breastfeeding for Mothers measured by structured questionnaire | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Salete de matos, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No